CLINICAL TRIAL: NCT02999022
Title: Lithium for Fracture Treatment: a Double Blind Randomized Controlled Trial
Brief Title: Lithium for Fracture Treatment: a Double Blind Randomized Controlled Trial (LiFT)
Acronym: LiFT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LiFT001
Record Dates: First submitted 2016-09-09; First posted 2016-12-21 (Estimated); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Fractures
Keywords: bone fractures; bony callus; fractures, bone; lithium; lithium carbonate; osteogenesis; bone development; fracture healing; fracture repair
MeSH Terms: conditions — Fractures, Bone; Callosities | interventions — Lithium Carbonate; Lithium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lithium carbonate (Experimental): Lithium carbonate 300mg capsule; once per day for 2 weeks.
  Interventions: Drug: Lithium Carbonate
- Lactose placebo (Placebo Comparator): Lactose placebo capsule; once per day for 2 weeks.
  Interventions: Drug: Lactose Placebo

INTERVENTIONS:
Drug: Lithium Carbonate — Intervention begins 14 days after injury for non-surgical participants and 2 weeks after surgery for participants who have surgical treatment of their fractures.
  Other Names: Lithium
  Arms: Lithium carbonate
Drug: Lactose Placebo — Intervention begins 14 days after injury for non-surgical participants and 2 weeks after surgery for participants who have surgical treatment of their fractures.
  Other Names: placebo
  Arms: Lactose placebo

SUMMARY:
This is a study designed to see if a low dose of Lithium treatment, taken for 2 weeks, can improve fracture healing and improve patients' function and productivity.

DETAILED DESCRIPTION:
Despite the success of traditional treatments for broken bones (surgery, immobilization, or both) 10% of fractures do not heal or take longer than normal to heal. This can have a significant effect on a patient's function and productivity, as well as on healthcare expenditures. Very few advances in fracture healing have been made, despite the need for new approaches to fracture treatment. This study proposes a simple, economical, and non-invasive approach to complement traditional fracture treatment that could decrease healing time and reduce the incidence of delayed healing. The investigators think that this can improve health outcomes for patients and reduce health care costs for the healthcare system in general. The goal is to see if a low-dose of Lithium treatment can have a positive effect on fracture healing and can reduce pain and improve function in patients who have broken a bone.

The LiFT study is a participant, surgeon and observer blinded single-centre randomized (1:1), controlled, superiority trial with 2 parallel groups. A minimization procedure will stratify participants based on the fractured long bone (clavicle, humerus, femur or tibia/fibula) and smoking.

Participants will be randomized to 1 of 2 groups: lithium capsules or placebo. The Lithium/placebo will be taken daily for 2 weeks, starting 2 weeks after the fracture occurs (or 2 weeks after surgery if the participant is treated with surgery).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55 years.
2. ASA (American Society of Anesthesiologists) ≤ 2 class (healthy) prior to injury.
3. Diaphyseal fracture of the humerus, femur or combined tibia/fibula (OTA diaphyseal subclass 2A or B), and clavicle (OTA diaphyseal subclass B1 or B2), with or without nerve injury.
4. Fracture that is primarily closed or open fracture that has complete wound coverage.
5. Randomization ≤14 days from injury or surgery (for surgical patients).
6. Fractures treated surgically or nonsurgically by endochondral/secondary bone healing.
7. For surgical patients, surgery must be within 14 days of injury.

Exclusion Criteria:

1. Currently pregnant or breastfeeding.
2. Any past or current malignancy that, in the opinion of an investigator, is not medically controlled.
3. Metabolic bone disease based on clinical history that, in the opinion of an investigator, is not medically controlled.
4. Autoimmune disease that, in the opinion of an investigator, is not medically controlled.
5. Hypothyroidism based on clinical history that, in the opinion of an investigator, is not medically controlled.
6. Renal impairment based on clinical history.
7. Past allergy or adverse reaction to Lithium.
8. Lactose intolerance.
9. Fractures surgically treated with absolute stability/primary bone healing.
10. Isolated tibia or isolated fibula fracture.
11. Currently taking Lithium or anti-psychotic or anti-seizure medication for the treatment of these conditions or at the discretion of an investigator.
12. Inability to comply with study protocol, in the opinion of the investigator(s).
13. Participation in another interventional clinical trial, at the discretion of the principal investigator.
14. Use of concomitant ultrasound or other bone stimulation device.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-07-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
radiographic healing of fracture | 8 weeks after injury (non-surgical participants) or 8 weeks after surgery (surgical participants)
  radiographic healing using the RUST score at 8 weeks

SECONDARY OUTCOMES:
radiographic union of fracture | 4, 6, 12, and 24 weeks after injury (non-surgical participants) or 4, 6, 12, and 24 weeks after surgery (surgical participants)
  time to radiographic union using the RUST score
visual analogue pain score | baseline then 4, 6, 8, 12, and 24 weeks after injury (non-surgical participants) or baseline then 4, 6, 8, 12, and 24 weeks after surgery (surgical participants)
  changes from baseline in participant-reported average pain in past week as measured on a visual analogue scale from 0-10 where 0 is no pain and 10 is extreme pain
physical function | baseline then 4, 6, 8, 12, and 24 weeks after injury (non-surgical participants) or baseline then 4, 6, 8, 12, and 24 weeks after surgery (surgical participants)
  changes in participant-reported function from baseline as measured on the RAND SF36 questionnaire
NSAID use | baseline then 3, 4, 6, 8, 12, and 24 weeks after injury (non-surgical participants) or baseline then 3, 4, 6, 8, 12, and 24 weeks after surgery (surgical participants)
  to track participant-reported use of non-steroidal anti-inflammatory medication and measure changes over the course of the study
re-operation (after initial fracture management) | 4, 6, 8, 12, and 24 weeks after injury (non-surgical participants) or 4, 6, 8, 12, and 24 weeks after surgery (surgical participants)
  surgery required after initial fracture management
adverse events | 2-6 weeks after injury (non-surgical participants) or 2-6 weeks after surgery (surgical participants)
  the number and type of adverse events occuring after the first dose of lithium/placebo and until the 6-week visit will be collected and reported according to local and national rules and regulations

CONTACTS AND LOCATIONS:
Overall Officials: Diane Nam, MSc,MD,FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (5):
- Canada (5):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario
  - The Ottawa Hospital Civic Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Unity Health St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nam D, Balasuberamaniam P, Milner K, Kunz M, Vachhani K, Kiss A, Whyne C. Lithium for Fracture Treatment (LiFT): a double-blind randomised control trial protocol. BMJ Open. 2020 Jan 7;10(1):e031545. doi: 10.1136/bmjopen-2019-031545. PMID 31915160